CLINICAL TRIAL: NCT06506006
Title: A Comparison of Early Outcome of Surgical Management of Proximal Humerus Fracture in Adults During COVID-19 Pandemic- A Prospective Cohort Study
Status: Completed | Type: Observational
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, ashbin bhattarai, Principal Investigator, B.P. Koirala Institute of Health Sciences
Other Study IDs: 306/077/078-IRC
Record Dates: First submitted 2024-07-16; First posted 2024-07-17 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Proximal Humerus Surgery in Covid Recovered Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- post COVID: patients with proximal humerus fracture with concommitant COVID postive status receiving delayed treatment
  Interventions: Biological: Covid infection
- Non COVIID: patients with proximal humerus fracture without concommitant COVID postive status receiving usual treatment
  Interventions: Biological: Covid infection

INTERVENTIONS:
Biological: Covid infection — outcome with and without covid infection

SUMMARY:
The goal of this observational study is to learn the outcome of proximal humerus fracture surgery in patients who had it delayed due to COVID infection and compare it with normal patients with same fracture and treatment. The main question it aims to answer is:

• Do the patients with proximal humerus fracture undergoing delayed fixation secondary to COVID infection have the same outcome as that of the normal patients?

The outcome of patients of both group will be assessed objectively via the standard Neer"s shoulder score and compared using independent variable T test.

ELIGIBILITY:
Inclusion Criteria:

* isolated traumatic proximal humerus fracture (Neer's grading 3 and 4)
* above 18 years of age
* consenting for the study

Exclusion Criteria:

* open fractures: Gustilo Grade II and III
* neurovascular compromise.
* neuromuscular disorders.
* injury severity score >16
* humerus fracture with extension to shaft

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: both group included patients with isolated traumatic proiximal humerus fracture. The post COVID group included patients with tested COVID positive at presentation. The Non COVID group wire non infected population without COVID infection
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
neer's shoulder score | 6 months
  functional scoring that includes combined score of range of motion, pain, function and anatomy, maximum score of 100 and minimum of 0 and higher score means better result

CONTACTS AND LOCATIONS:
Overall Officials: ashbin bhattarai, masters, Principal Investigator — National Trauma Center
Locations (1):
- B.P.Koirala Insitute of Helath Sciences, Dharān, Koshi, Nepal

IPD SHARING:
Plan to Share IPD: No
only the results will be shared which includes the mean score and p values between groups